CLINICAL TRIAL: NCT05396261
Title: Post-marketing Surveillance of a Flexible Wound Dressing for the Management of Genital Skin Conditions
Brief Title: a Flexible Wound Dressing for the Management of Genital Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stratpharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPASMSX01 HALL
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Vaginitis; Atrophic Vaginitis; Lichen Planus; Lichen Sclerosus; Menopause Related Conditions
MeSH Terms: conditions — Vaginitis; Atrophic Vaginitis; Lichen Planus; Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Film forming silicone gel (7-0940) is an innovative gel that forms a full contact, flexible wound dressing for supporting mucosal conditions of the genital, rectal and perineal areas.
  Film forming silicone gel (7-0940) is a semi-occlusive, non-resorbable, self-drying and transparent gel.
  Film forming silicone gel (7-0940) may be directly applied to dry, wet, cracked and sensitive mucosal tissue.
  Film forming silicone gel (7-0940) gel is bacteriostatic and inert. It contains no alcohols, parabens or fragrances.
  Interventions: Device: Film forming silicone gel (7-0940)

INTERVENTIONS:
Device: Film forming silicone gel (7-0940) — Anecdotal evidence suggests that genital conditions in women associated with vaginal atrophy improve with the use of film-forming silicone dressings.

SUMMARY:
The objective of the study is to determine the efficacy of 7-0940 in the management of genital skin conditions in female patients

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Diagnosed genital skin condition

Exclusion Criteria:

* Unable to give informed consent
* Patient unable to apply topical device
* Allergy or intolerance to ingredients or excipients of the formulation of studied products

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
gynaecological skin condition | Duration of the therapy will be according to physician's clinical practice. The average is 3 visits over a period of 3 to 6 months
  Likert scales to measure:
  * Dryness
  * Tissue thinning
  * Erosion/Ulcers
  * Fissures
  * Erythema
  * Scarring/adhesion
  * Contact bleeding
  * Bloodblisters
  * Greyish film
  * White lacy streaks

SECONDARY OUTCOMES:
patient symptoms | Duration of the therapy will be according to physician's clinical practice. The average is 3 visits over a period of 3 to 6 months
  Likert scales to measure:
  * Pruritus/itchiness
  * Tender/sore
  * Swelling
  * Dryness
  * Burning of skin
  * Dyspareunia
  * Stinging with urination/clothes
  * Defecating pain/burning

CONTACTS AND LOCATIONS:
Overall Officials: Philip Hall, MD, Principal Investigator — St. Andrews War Memorial Hospital - Australia
Locations (1):
- St. Andrews War Memorial Hospital, Spring Hill, Queensland, Australia

REFERENCES:
- [Derived] Hall P. A Feasibility Study Investigating a Topical Preparation as Novel Adjunct Treatment for the Symptomatic Management of Vulvovaginal Skin Conditions. Womens Health Rep (New Rochelle). 2024 May 17;5(1):444-452. doi: 10.1089/whr.2024.0026. eCollection 2024. PMID 39035147